CLINICAL TRIAL: NCT00178204
Title: Sleep Architecture and Chemotherapy-Related Fatigue
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Joseph Roscoe, Research Associate Professor, University of Rochester
Other Study IDs: MRSG-04-233-01-CPPB
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Fatigue; Sleep; Cancer
Keywords: delta sleep; Cancer-related fatigue; Sleep Disturbance; chemotherapy
MeSH Terms: conditions — Fatigue; Neoplasms; Parasomnias

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify specific chemotherapy-related changes in sleep stages/architecture that may relate to an increase in fatigue in individuals with cancer.

The researchers hypothesize that the fatigue experienced by cancer patients receiving chemotherapy is in part due to changes in restorative sleeping during the non-rapid eye movement cycles of sleep (i.e., delta activity).

DETAILED DESCRIPTION:
Studies have shown a strong positive correlation between self-reported changes in sleep and cancer patients' fatigue, and also between an objective measure of sleep continuity, [i.e., actigraphy and polysomnography (PSG)] and self-reported fatigue. Chemotherapy disrupts normal sleep patterns, and fatigue, in the later stages of chemotherapy, may occur as a result of disturbed nocturnal sleep continuity. However, the causes of chemotherapy-related fatigue remain unknown, and whether or not abnormal sleep architecture contributes to this debilitating effect has yet to be explored. We believe that fatigue experienced by many cancer patients receiving chemotherapy is due, at least in part, to changes in delta activity [i.e., restorative sleep during the non-rapid eye movement (NREM) cycles of sleep]. A finding that slow wave sleep abnormalities play a significant role in fatigue would prompt further confirmatory studies and support controlled intervention studies.

Comparisons: In a clinical trial of individuals with cancer prior to, during, and after completion of chemotherapy, we will identify and compare specific chemotherapy-related changes in sleep stages/architecture that may relate to an increase in fatigue. These changes will be measured by actigraphy, PSG, and patient self-reporting techniques (e.g., sleep diaries, questionnaires).

The primary objective is to:

* examine the role of delta sleep in the development of chemotherapy-induced fatigue in cancer patients

Secondary objectives are to:

* characterize the involvement of other elements of sleep architecture [e.g., rapid eye movement (REM) sleep] and changes in sleep continuity relating to the development of chemotherapy-induced fatigue in cancer patients
* examine the role of sleep architecture in the persistence of chemotherapy-induced fatigue
* examine (in post hoc analyses) the relationship of various physical symptoms and patient variables that may be related to fatigue (e.g., pain, hot flashes, anxiety, hemoglobin, menopausal status, sleep continuity, and QOL) and to each other, both during and following chemotherapy.

Answers to these questions will provide information that will be helpful in developing potential targets for interventions to reduce fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of cancer and not have had chemotherapy during the prior three years
* Be scheduled for chemotherapy that is expected to last at least 9 weeks but not more than 33 weeks without concurrent interferon treatment. Radiation therapy is allowed provided it is concluded within the 33 week time period
* Have a stable sleep/wake schedule (no shift work) with a preferred sleep phase between 10:00 PM and 9:00 AM
* Be 18 years of age or older
* Give informed consent
* If on beta blockers or being treated for depression or a thyroid disorder, the medication has been stable for 3 months

Exclusion Criteria:

* On a short term basis (less than 3 months), taking any prescription medication for the control of anxiety, sleep, depression, or fatigue OR taking any over-the-counter medications known to affect sleep
* Diagnosed with post-traumatic stress disorder (PTSD) or have a substance abuse disorder or psychotic disorder (currently or by history)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients beginning chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2004-11; Primary Completion 2009-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Polysomnography (PSG) | Two consecutive nights prior to first chemotherapy, approximately three weeks following the patient's last chemotherapy, and three months following the last treatment.
  Polysomnography provides direct and quantitative measures of cortical activity during sleep (in the form of brain waves). The sleep continuity data derived from this technique include sleep latency (time taken to fall asleep), wake after sleep onset time, total sleep time, and sleep efficiency (SE). The sleep architecture information derived from this technique consists of the assessment of sleep in terms of its constituent component stages (i.e., percent Stage-1, Stage-2, SWS, and REM sleep).

SECONDARY OUTCOMES:
Brief Fatigue Inventory (BFI) | On the first night of each of the three polysomnography assessments
  The Brief Fatigue Inventory is a 9-item, patient-report instrument with established reliability and validity that allows for the rapid assessment of fatigue level in cancer patients. Possible scores on this scale range from 0 - 10 with higher numbers indicating greater fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Joesph A Roscoe, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester James P. Wilmot Cancer Center, Rochester, New York, United States